CLINICAL TRIAL: NCT06760182
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of TQH2722 Injection Combined With Background Therapy in Patients With Seasonal Allergic Rhinitis
Brief Title: Clinical Trial of TQH2722 Injection in Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH2722-II-05
Record Dates: First submitted 2024-12-25; First posted 2025-01-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQH2722 injection (Experimental)
  Interventions: Drug: TQH2722 injection
- TQH2722 Placebo (Placebo Comparator): TQH2722 placebo, 1 weeks as a treatment cycle.
  Interventions: Drug: TQH2722 Placebo

INTERVENTIONS:
Drug: TQH2722 injection — TQH2722 injection is a humanized monoclonal antibody targeting interleukin-4 receptor alpha (IL-4Rα).
  Arms: TQH2722 injection
Drug: TQH2722 Placebo — Placebo without drug substance.
  Arms: TQH2722 Placebo

SUMMARY:
To evaluate TQH2722 injection in all patients receiving background treatment with mometasone furoate nasal spray (MFNS) and loratadine. The efficacy, safety and immunogenicity of the solution in patients with seasonal allergic rhinitis compared with placebo are expected to include 168 patients with confirmed seasonal allergic rhinitis (SAR) who have failed to respond to standard treatments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years at the screening period.
* Patients who met the diagnostic criteria of allergic rhinitis in Chinese Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (revised edition, 2022)
* Positive of at least 1 allergen skin prick test(SPT) and/or serum-specific IgE within 1 year before enrollment.
* Subjects have sufficient pollen exposure during the pollen season:
* Subjects' medical history suggested that SAR symptoms were poorly controlled or subjects' subjective symptoms were not satisfactorily controlled after drug treatment during the same pollen season in the past.
* On the day of screening, the iTNSS score in the morning was ≥4; At baseline visit, the morning iTNSS was ≥4 points, and the average score of the past 6 rTNSS was ≥6 points;
* At baseline visit, the absolute value of peripheral blood eosinophils was ≥0.15×109/L;
* During the screening/induction period, the subjects had good compliance;
* Subjects with asthma who were assessed by the investigator or specialist as having stable asthma;
* Voluntary participation in this trial and signing the informed consent form
* Subjects (including partners) have no pregnancy and voluntarily take one or more non-pharmaceutical measures for contraception at period from drug administration to 6 months after the last study drug administration

Exclusion Criteria:

* Laboratory test values did not meet the requirements during screening or randomization
* Any disease that the investigator believes interferes with the patient's ability to complete the entire course of the study;
* Patients with active autoimmune disease
* People with known or suspected immunosuppression
* Subjects with active malignancy or a history of malignancy;
* Active hepatitis or hepatitis B was present during the screening period; Or human immunodeficiency virus antibody (Anti-HIV) positive, or treponema pallidum antibody (Anti-TP) positive;
* Diagnosis of helminthic infection within 6 months prior to screening, not receiving standard treatment or not responding to standard treatment;
* Subjects who have undergone nasal surgery or sinus surgery within 6 months before screening
* Subjects have concomitant medical conditions that preclude them from completing the screening period assessment or evaluating the primary efficacy endpoint;
* Subjects with nasal malignancies and benign tumors;
* History of hypersensitivity to any content of the study drugs or its excipients
* Subjects with a history of systemic allergy to any biological agent;
* Pregnant or lactating women;
* Alcohol, drug and known drug dependence;
* Have a history of vital organ transplantation or hematopoietic stem cell/bone marrow transplantation;
* Any medical or psychiatric condition that, in the investigator's judgment, puts the subject at risk, interferes with participation in the study, or interferes with the interpretation of the study results;
* Any condition that the investigator or primary physician believes may not be appropriate for participating the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Retrospective nasal symptom score after treatment for 2 weeks | Baseline up to 2 weeks
  Average daily retrospective nasal symptom score (rTNSS) changed from baseline after 2 weeks of treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.

SECONDARY OUTCOMES:
Retrospective nasal symptom score after treatment for 4 weeks | Baseline up to 4 weeks
  Mean daily retrospective nasal symptom total score (rTNSS) changes from baseline at 4 weeks of treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Mean daily changes in retrospective nasal symptom total score | Baseline up to 2 and 4 weeks
  Mean daily changes in retrospective nasal symptom total score (AM rTNSS) from baseline at 2 weeks and 4 weeks after treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Mean daily nightly retrospective nasal symptom total score | Baseline up to 2 and 4 weeks
  Mean daily nightly retrospective nasal symptom total score (PM rTNSS) changes from baseline at 2 weeks and 4 weeks after treatment. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Instantaneous nasal symptom score: Mean change of instantaneous nasal symptom total score (iTNSS) from baseline | Baseline up to 2 and 4 weeks
  Mean change of instantaneous nasal symptom total score (iTNSS) from baseline every morning before treatment for 2 weeks and 4 weeks. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Instantaneous nasal symptom score: Mean daily rTNSS change from baseline | Baseline up to 2 and 4 weeks
  Mean daily rTNSSchange from baseline at 2 weeks and 4 weeks of treatment; The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Instantaneous nasal symptom score: Mean change rate of iTNSS from baseline | Baseline up to 2 and 4 weeks
  Mean change rate of iTNSS from baseline before treatment at 2 weeks and 4 weeks each morning. The total score is 0-12 points, with the higher score meaning the more severe symptoms.
Instantaneous nasal single symptom score: Mean changes from baseline in daily retrospective nasal symptom scores | Baseline up to 2 and 4 weeks
  Mean changes from baseline in daily retrospective nasal symptom scores (runny nose, nasal congestion, nasal itchy, and sneezing) at 2 and 4 weeks of treatment. The single score is 0-3 points, with the higher score meaning the more severe symptoms.
Instantaneous nasal single symptom score: Mean changes from baseline in scores of individual nasal symptoms during the day | Baseline up to 2 and 4 weeks
  Mean changes from baseline in scores of individual nasal symptoms (runny nose, nasal congestion, itchy nose, and sneezing) were reviewed daily (AM) at 2 weeks and 4 weeks of treatment. The single score is 0-3 points, with the higher score meaning the more severe symptoms.
Instantaneous nasal single symptom score: Mean changes from baseline in scores of individual nasal symptoms at night | Baseline up to 2 and 4 weeks
  Mean changes from baseline in scores of individual nasal symptoms (runny nose, nasal congestion, nasal itchy and sneezing) at night (PM) after 2 and 4 weeks of treatment. The single score is 0-3 points, with the higher score meaning the more severe symptoms.
Retrospective ocular symptom score: Mean changes in daily retrospective ocular symptom score | Baseline up to 2 and 4 weeks
  Mean changes in daily retrospective ocular symptom score (rTOSS) from baseline at 2 and 4 weeks of treatment; The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Retrospective ocular symptom score: Mean changes in retrospective ocular symptom score during the day | Baseline up to 2 and 4 weeks
  Mean daily changes in retrospective ocular symptom score (AM rTOSS) from baseline at 2 weeks and 4 weeks of treatment. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Retrospective ocular symptom score: Mean retrospective ocular symptom score at night | Baseline up to 2 and 4 weeks
  Mean nightly retrospective ocular symptom score (PM rTOSS) changes from baseline at 2 weeks and 4 weeks of treatment. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Retrospective ocular symptom score: Mean change of instantaneous ocular symptom total score | Baseline up to 2 and 4 weeks
  Mean change of instantaneous ocular symptom total score (iTOSS) from baseline every morning at 2 weeks and 4 weeks of treatment. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Retrospective ocular symptom score: Mean rate of change in daily rTOSS | Baseline up to 2 and 4 weeks
  Mean rate of change in daily rTOSS from baseline at 2 and 4 weeks of treatment. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Retrospective nasal symptom score: Average daily retrospective nasal symptom score | Baseline up to 4 weeks
  Average daily retrospective nasal symptom score (rTNSS) changed from baseline after 4 weeks of treatment. The total score is 0-12points, with the higher score meaning the more severe symptoms.
Retrospective ocular symptom score: Mean change rate of iTOSS each morning | Baseline up to 2 and 4 weeks
  Mean change rate of iTOSS from baseline before treatment at 2 weeks and 4 weeks each morning. The total score is 0-9 points, with the higher score meaning the more severe symptoms.
Instantaneous ocular single symptom score: Average changes in scores of individual ocular symptoms | Baseline up to 2 and 4 weeks
  Average changes in scores of individual ocular symptoms (itchy, tearing, red eyes) at 2 and 4 weeks of treatment compared with baseline. The single score is 0-3 points, with the higher score meaning the more severe symptoms
Instantaneous ocular single symptom score: Average changes of individual ocular symptom scores during the day | Baseline up to 2 and 4 weeks
  Average changes of individual ocular symptom scores (itchy, watery eyes, red eyes) compared with baseline were reviewed daily (AM) at 2 weeks and 4 weeks of treatment. The single score is 0-3 points, with the higher score meaning the more severe symptoms.
Instantaneous ocular single symptom score: Average changes of individual ocular symptoms at night | Baseline up to 2 and 4 weeks
  Average changes of individual ocular symptoms (itchy, watery eyes, red eyes) scores at night (PM) after 2 weeks of treatment and 4 weeks of treatment compared with baseline. The single score is 0-3 points, with the higher score meaning the more severe symptoms.
Quality of life questionnaire | Baseline up to 2 and 4 weeks
  Changes in quality of life questionnaire (RQLQ) scores from baseline for patients with allergic rhinitis after 2 weeks and 4 weeks of treatment. The total score is 0-168 points, with the higher score meaning the more severe symptoms.
Time of onset | Baseline up to 4 weeks
  Time of onset after treatment.
Time to Reach Maximum Plasma Concentration (Tmax) | Baseline up to 4 weeks
  Time to reach maximum plasma concentration after administration.
Area under the curve | Baseline up to 2 and 4 weeks
  Area under the curve of mean daily rTNSS change from baseline at 2 and 4 weeks of treatment
Number of days with no or mild symptoms of Allergic rhinitis symptoms | Baseline up to 2 and 4 weeks
  Number of days with no or mild symptoms during 2 weeks and 4 weeks of treatment
Adverse event rate | Baseline up to 12 weeks
  Incidence and severity of adverse events (AE) and serious adverse events (SAE), physical examination, vital signs, 12-lead electrocardiogram (ECG), and abnormal laboratory indicators.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of science and technology, Wuhan, Hubei
  - Tongji Hospital of Tongji medical college of HUST, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Ansteel Group General hospital, Anshan, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Health Industry Group Iron Coal General Hospital, Tieling, Liaoning
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Second Provincial General Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Qilu, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan